CLINICAL TRIAL: NCT05141734
Title: Evaluation of Patients With Benign Paroxysmal Positional Vertigo With vHIT (Video Head Impulse Test) and VNG (Videonystagmography)
Brief Title: Correlation Tests for Patients With Benign Paroxysmal Positional Vertigo
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Selcuk University Faculty of Medicine, Selcuk University
Other Study IDs: 2019/54
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Positional Vertigo; Reflexes, Vestibo-Ocular; Nystagmus Vestibular
Keywords: vestibular function tests; Head Impulse Test; semicircular canals
MeSH Terms: conditions — Vertigo | interventions — Reflex, Vestibulo-Ocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPPV (benign paroxysmal positional vertigo): VOR gains were measured by vHIT in both the study group and the control group. The SPV values of the nystagmus observed during the Dix-Hallpike maneuver in the study group were recorded by Videonystagmography (VNG) and compared with the VOR gains.
  Interventions: Diagnostic Test: The relationship between the vestibulo-ocular reflex (VOR) gains and the slow phase velocity (SPV)
- Control: VOR gains were measured by vHIT in both the study group and the control group. The SPV values of the nystagmus observed during the Dix-Hallpike maneuver in the study group were recorded by Videonystagmography (VNG) and compared with the VOR gains.
  Interventions: Diagnostic Test: The relationship between the vestibulo-ocular reflex (VOR) gains and the slow phase velocity (SPV)

INTERVENTIONS:
Diagnostic Test: The relationship between the vestibulo-ocular reflex (VOR) gains and the slow phase velocity (SPV) — The vestibulo-ocular reflex (VOR) gains were measured by video Head Impulse Test (vHIT) in both the study group and the control group. The slow phase velocity (SPV) values of the nystagmus observed during the Dix-Hallpike maneuver in the study group were recorded by Videonystagmography (VNG) and compared with the VOR gains.

SUMMARY:
This study aimed to investigate whether there is a relationship between nystagmus intensity and vestibular-ocular reflex gains by comparing Videonystagmography and video head impulse test in patients with posterior semicircular canal-benign paroxysmal positional vertigo.

DETAILED DESCRIPTION:
The aim of this study is to investigate the relationship between the vestibulo-ocular reflex (VOR) gains obtained by video Head Impulse Test (vHIT) and the slow phase velocity (SPV) of nystagmus in patients with benign paroxysmal positional vertigo (BPPV) originating from the posterior semicircular canal (PSCC).

The patients were included in two groups. The study group consisted of patients with isolated PSCC BPPV (PSCC-BPPV), and the control group consisted of age and gender-matched healthy individuals. VOR gains were measured by vHIT in both the study group and the control group. The SPV values of the nystagmus observed during the Dix-Hallpike maneuver in the study group were recorded by Videonystagmography (VNG) and compared with the VOR gains.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated benign paroxysmal positional vertigo were included in the study group.
* The patients included in the control group were composed of those who did not complain of vertigo.

Exclusion Criteria:

-Participants with a history of neuro-otologic disease, an orthopedic disease that prevents neck movements, and any disease or surgery that causes impairment in ocular movements were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients included in the study group were diagnosed with isolated benign paroxysmal positional vertigo (BPPV) according to clinical symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Comparison of nystagmus intensity and vestibulo-ocular reflex gains in patients with benign paroxysmal positional vertigo | 2019-2010 (15 months)
  The vestibulo-ocular reflex (VOR) gains and the slow phase velocity (SPV) of nystagmus were compared in patients with benign paroxysmal positional vertigo.

CONTACTS AND LOCATIONS:
Overall Officials: Merih Onal, MD, Principal Investigator — Selcuk University
Locations (1):
- Merih Onal, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Onal M, Aygun A, Colpan B, Karakayaoglu H, Onal O. Correlation between nystagmus intensity and vestibular-ocular reflex gain in benign paroxysmal positional vertigo: A prospective, clinical study. J Vestib Res. 2023;33(2):115-125. doi: 10.3233/VES-220106. PMID 36776086